CLINICAL TRIAL: NCT00598650
Title: A Long-term, Extension Study of E2020 in Patients With Dementia With Lewy Bodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020-J081-432
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Dementia With Lewy Bodies (DLB)
Keywords: Lewy Body Disease; Dementia; Clinical Trial; Phase II; E2020; donepezil hydrochloride
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — Donepezil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E2020

INTERVENTIONS:
Drug: E2020 — Dosage and administration: Patients will receive oral administration of 1 tablet of 3 mg (E2020) from Day 1 to Day 14 of treatment period, 1 tablet of 5 mg (E2020) from Day 15 onwards once daily after breakfast.
  Other Names: Aricept

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of E2020 in patients with Dementia with Lewy Bodies (DLB).

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed as probable Dementia with Lewy Bodies (DLB) according to the diagnostic criteria for DLB.
2. Patients who have completed Phase II double-blind study (E2020-J081-431).
3. Patients having caregivers who submit written consent for cooperative involvement in this study, can routinely stay with patients 3 days a week (at least 4 hours a day), provide patients' information necessary for this study, assist treatment compliance and escort their patients on required visits to study institution.

Exclusion criteria:

1. Patients with a complication of serious neuropsychiatric disease(s) such as stroke, brain tumor, schizophrenia, epilepsy, normal pressure hydrocephalus, mental retardation, brain trauma with unconsciousness, and/or who underwent brain surgery causing unsolved deficiency.
2. Patients with severe complication of cardiovascular, hepatic, renal, hematological, or other diseases unable to secure the safety.
3. Pregnant or lactating women, or women who are willing to become pregnant no later than 1 month after the scheduled study completion.
4. Patients with severe extrapyramidal disorders (Hoehn and Yahr staging score is greater than IV).
5. Patients whose systolic blood pressure is less than 90 mmHg or pulse rate is less than 50 beats/min.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itaru Arimoto, Study Director — New Product Development, Clinical Research Center, Eisai Co., Ltd.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E2020
Started | 108
Completed | 81 (5 subjects withdrew for multiple reasons)
Not Completed | 27
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 18
Not completed — No treatment for 3 weeks | 1
Not completed — Not eligible | 1
Not completed — Prohibited Concomitant Medication | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | E2020
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 40
Weight [Mean (Standard Deviation); unit: kg] | 49 (9.24)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mini-mental State Examination (MMSE) Total
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranged from 0 - 30, where a higher score indicated better cognitive state.
Time Frame: Baseline, Week 52, and Week 52 LOCF
Population: Efficacy Analysis Set: subjects who received at least one dose of E2020 and also provided safety assessment data after baseline, with at least one available efficacy evaluation. Two subjects whose diagnosis was suspected not to meet clinical criteria of probable DLB and 2 subjects with lack of efficacy data were excluded from the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Placebo/E2020: Of the 104 patients of Arm 1, Arm 2 is patients from the placebo group in the preceding a 12-week, randomized, placebo-controlled trial (registered at ClinicalTrials.gov, number NCT00543855). That is to say Arm 1 consisted of 28 patients (Arm 2) from the placebo group in the preceding trial, and 76 patients from any of the E2020 group (3-mg group, 5-mg group, or 10-mg group).
Arm/Group | E2020 | Placebo/E2020
Number analyzed (Participants) | 104 | 28
Score on a Scale
  Baseline | 20.9 (5.1) | 18.6 (4.7)
  Week 52 | 0.3 (3.7) | 2 (4.4)
  Week 52 LOCF | 0.2 (3.5) | 1.7 (4.4)

2. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Score of Psychiatric Symptoms
Description: NPI measured 10 different domains of psychiatric symptoms including delusion and hallucination. Each domain is scored for: present or absent, frequency, and severity. The score derived from sub-scores; total ranged from "0" to "120," higher score indicated worse neuropsychiatric outcomes.
Time Frame: Baseline, Week 52, and Week 52 LOCF
Population: Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | E2020 | Placebo/E2020
Number analyzed (Participants) | 104 | 28
Score on a Scale
  Baseline | 13.1 (16.8) | 17.8 (8.2)
  Week 52 | -1.9 (9.8) | -4.1 (10.1)
  Week 52 LOCF | -0.7 (11.1) | -4.3 (9.7)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: Other adverse events are listed at a frequency of 5% or greater
Arm/Group | E2020
Serious Adverse Events (participants affected / at risk) | 8/108
Other Adverse Events (participants affected / at risk) | 53/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E2020 (N=108)
Compression fracture (Injury, poisoning and procedural complications) | 3
Psychiatric symptom (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Poriomania (Psychiatric disorders) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar infarction (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 3
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Gastrointestinal mucosal exfoliation (Gastrointestinal disorders) | 1
Radial nerve palsy (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myocardial infarction (Cardiac disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Pseudomembranous colitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E2020 (N=108)
Nasopharyngitis (Infections and infestations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 6
Insomnia (Psychiatric disorders) | 6
Parkinsonism (Nervous system disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 8
Blood creatine phosphokinase increased (Investigations) | 12
Blood pressure increased (Investigations) | 11
Blood urine present (Investigations) | 7
Protein urine present (Investigations) | 7
Contusion (Injury, poisoning and procedural complications) | 12
Fall (Injury, poisoning and procedural complications) | 11
Compression fracture (Injury, poisoning and procedural complications) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other